CLINICAL TRIAL: NCT03509506
Title: Usability and Effectiveness of a Self-care Mobile Health App in Individuals With Heart Failure
Brief Title: A Self-care Mobile Health App in Individuals With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19985
Record Dates: First submitted 2018-04-09; First posted 2018-04-26 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Self-Management; Mobile Applications; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-App Group (No Intervention): The participants will be instructed to continue their daily routine, track their daily steps with a pedometer, and record their daily steps on the "Activity Log" paper form.
- App Group (Experimental): The participants will be trained how to use the mobile application (Heart Failure Health Storyline (HFHS)) to track their health status, physical activity, manage their medications schedule, and explore the other features that the application has. Additionally, they will receive a pedometer to track their daily steps and record their data on the mobile application.
  Interventions: Behavioral: App Group

INTERVENTIONS:
Behavioral: App Group — The participants will be educated to use the HFHS application to monitor their daily vital signs (HR, BP, body weight), physical activity, and medications for 4 weeks.
  The research team will monitor their data entry remotely via the HFHS App. The team will text the participant via the App if one or more of following conditions is noted:
  * The vital signs show undesired readings
  * The records on the HFHS App show that the participant did not take the medications as the schedule says
  In addition, the team will call the participant 3 days later to follow up regarding the participant's action towards the text message that the team sent.
  Arms: App Group

SUMMARY:
This study was designed to determine the potential benefits that individuals with heart failure (HF) could experience from using a mobile application.

DETAILED DESCRIPTION:
The mobile application is called the Heart Failure Health Storylines (HFHS). The potential benefits will be examined by determining the changes in physical activity and quality of life of the participants, who will use the application and compare the results with the participants, who will not use the application.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic heart failure, class I - III based on New York Heart Association (NYHA) scale
* Walking independently with/without an assistive device

Exclusion Criteria: The participant will be excluded if one or more of the following is present

* Cognitive impairment (< 26 on Montreal Cognitive Assessment).
* Uncorrected vision
* Hearing problems
* Neurological disorders.
* Cannot speak and read the English language,
* Not owning a smart cell phone with internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Quality of Experience | Change from baseline to 4 weeks
  The Quality of Experience (QoE) survey will be used to measure the quality of experience in using the mobile application

SECONDARY OUTCOMES:
Quality of Life for Individuals with Heart Failure | Change from baseline to 4 weeks
  36-Item Short-Form Health Survey (SF-36 version 1.0)
Quality of Life for Individuals with HF | Change from baseline to 4 weeks
  Minnesota Living with Heart Failure (MLHF) questionnaire
Physical Activity will be indicated by daily step counts | Change from baseline to 4 weeks
  Physical activity will be assessed with a pedometer

CONTACTS AND LOCATIONS:
Overall Officials: Suh Jen Lin, PhD, PT, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States